CLINICAL TRIAL: NCT02929186
Title: Opt-In Versus Opt-Out for Colorectal Cancer Screening Outreach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 826047
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Cancer of the Colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opt-In (Experimental): Opt-In Outreach
  Interventions: Behavioral: Opt-In Outreach
- Opt-Out (Experimental): Opt-Out Outreach
  Interventions: Behavioral: Opt-Out Outreach

INTERVENTIONS:
Behavioral: Opt-In Outreach — Subjects will receive a communication (mail or electronic) describing the importance of colorectal cancer screening with the option to elect to receive a home FIT kit or report prior screening.
  Arms: Opt-In
Behavioral: Opt-Out Outreach — Subjects will receive a communication (mail or electronic) describing the importance of colorectal cancer screening with the option to choose not to receive a home FIT kit or report prior screening. A FIT kit will otherwise be sent to the subject as a default.
  Arms: Opt-Out

SUMMARY:
This is a randomized controlled pilot study aimed at testing different outreach strategies (opt-in versus opt-out) to increase colorectal cancer screening through completion of mailed home fecal immunohistochemical testing (FIT).

DETAILED DESCRIPTION:
This is a randomized controlled pilot study aimed at testing different outreach strategies to increase colorectal cancer screening using mailed fecal immunohistochemical testing (FIT). The investigators will randomize a cohort of subjects between the ages of 50-74 into 2 arms:

1. Opt-In - subject must actively choose to receive a home FIT kit.
2. Opt-Out - a FIT kit is sent as a default unless the subject actives chooses not to receive the kit or reports prior screening.

ELIGIBILITY:
Inclusion Criteria:

* Between 50 to 74 years old
* Has received care at the Division of Internal Medicine
* Due for screening
* Asymptomatic for colorectal cancer (CRC)

Exclusion Criteria:

* Has had prior colonoscopy within 10 years, sigmoidoscopy within 5 years, and fecal occult blood test (FOBT)/FIT within twelve months of the chart review (We will exclude patients who self-report undergoing any of the above procedures)
* Has a history of CRC
* Has a history of other GI cancer
* Has history of confirmed Inflammatory Bowel Disease (IBD) (e.g. Crohn's disease, ulcerative colitis; Irritable bowel syndrome does not exclude patients)
* Has history of colitis other than Crohn's disease or ulcerative colitis
* Has had a colectomy
* Has a relative that has been diagnosed with CRC
* Has been diagnosed with Lynch Syndrome (i.e. HNPCC)
* Has been diagnosed with Familial Adenomatous Polyposis (FAP)
* Has iron deficiency anemia
* Has history of lower GI bleeding
* Has metastatic (Stage IV) blood or solid tumor cancer
* Has end stage renal disease
* Has cirrhosis
* Has heart failure
* Has dementia
* Has any other condition that, in the opinion of the investigator, excludes the patient from participating in this study

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
FIT Completion Rate | 3 months
  The percentage of participants who successfully complete the FIT.

SECONDARY OUTCOMES:
Mail/Electronic Message Engagement | 3 months
  The percentage of people who send responses using either mail or electronic messaging.

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania; Chyke Doubeni, MD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No